CLINICAL TRIAL: NCT01776112
Title: Enhancing Synaptic Plasticity and Cognition by Physical Exercise and Cognitive Training in Schizophrenia: A Randomised Controlled Trial
Brief Title: Enhancing Synaptic Plasticity and Cognition in Schizophrenia
Acronym: EXERCISE-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Peter Falkai, Prof. Dr. med. Peter Falkai, University Medical Center Goettingen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMCG-EX-II
Record Dates: First submitted 2012-01-01; First posted 2013-01-25 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Schizophrenia
Keywords: schizophrenia; negative symptoms; cognitive deficits; synaptic plasticity
MeSH Terms: conditions — Schizophrenia; Cognition Disorders | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- SZ-Exercise (Experimental): Standard treatment and participation in the sports program (cycling) including cognitive training, 3 sessions cycling (30 min. each) per week for 3 months and 2 sessions Cogpack per week for the last 6 weeks.
  Interventions: Other: Exercise
- SZ-TableSoccer (Placebo Comparator): Standard treatment and participation in an activity without physical improvement as placebo condition (table soccer in groups of 4), but including cognitive training, 3 sessions (30 min. each) per week for 3 months and 2 sessions Cogpack per week for the last 6 weeks.
  Interventions: Other: TableSoccer
- HC-Exercise (Experimental): Standard treatment and participation in an activity without physical improvement as placebo condition (table football in groups of 4), but including cognitive training, 3 sessions (30 min. each) per week for 3 months and 2 sessions Cogpack per week for the last 6 weeks.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Standard treatment and participation in the sports program (cycling) including cognitive training, 3 sessions cycling (30 min. each) per week for 3 months and 2 sessions Cogpack per week for the last 6 weeks.
  Arms: HC-Exercise; SZ-Exercise
Other: TableSoccer — Standard treatment and participation in an activity without physical improvement as placebo condition (table football in groups of 4), but including cognitive training, 3 sessions (30 min. each) per week for 3 months and 2 sessions Cogpack per week for the last 6 weeks.
  Arms: SZ-TableSoccer

SUMMARY:
To explore: (a) if physical exercise (sports) combined with cognitive training leads to (superior) improvement of cognition in schizophrenia compared to sports or cognitive training alone (b) if a sports program alone or in combination with cognitive training has influence on hippocampal pathology and synaptic plasticity in schizophrenia compared to a placebo condition.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with the diagnosis of schizophrenia (based on ICD-10 criteria)
* Age between 18 and 55
* Verbal IQ ≥ 85
* Stable psychopathology on constant medication for 2 weeks
* Informed consent.

Exclusion Criteria:

Patients, who are

* not willing or able to participate in the sports program and cognitive training
* reveal a significant worsening of psychopathology (based on an increase over 20% of the PANSS positive score)
* have an organic mental disorder (such as intoxication or neurological disorders of the CNS)
* suffer from instable somatic diseases
* have an active substance abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2011-01; Primary Completion 2014-03 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Hippocampal volume | after three months of exercise
  Measurement of hippocampal volume before and after the exercise intervention, 3T-MRI MPRAGE-Sequence, manual and automated delineation of hippocampal borders

SECONDARY OUTCOMES:
Verbal Learning Memory | after three months of exercise
  Neuropsychological assessment of a working memory domain via the Verbal Learning Memory Test (German: Helmstaedter, C., Lendt, M., Lux, S., 2001. Verbaler Lern- und Merkfähigkeitstest (VLMT). Göttingen, Beltz)
Positive and negative symptoms | after three months of exercise
  Measurement of positive and negative symptoms of schizophrenia using the "Positive and Negative Symptom Scale for Schizophrenia" (Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Falkai, MD, PhD, Principal Investigator — Head, Dept. of Psychiatry and Psychotherapy University Medical Center Goettingen Georg-August-University von-Siebold-Strasse 5 D-37075 Goettingen Germany P: +49-(0)551-39-6610; Andrea Schmitt, MD, PhD, Study Director — Professor, Dept. of Psychiatry and Psychotherapy University Medical Center Goettingen Georg-August-University von-Siebold-Strasse 5 D-37075 Goettingen Germany P: +49-(0)551-39-6610; Berend Malchow, MD, Study Director — Senior Consultant, Dept. of Psychiatry and Psychotherapy University Medical Center Goettingen Georg-August-University von-Siebold-Strasse 5 D-37075 Goettingen Germany P: +49-(0)551-39-6610
Locations (1):
- Dept. of Psychiatry and Psychotherapy, University Medical Center Goettingen, Georg-August-University, Göttingen, Lower Saxony, Germany

REFERENCES:
- [Background] Pajonk FG, Wobrock T, Gruber O, Scherk H, Berner D, Kaizl I, Kierer A, Muller S, Oest M, Meyer T, Backens M, Schneider-Axmann T, Thornton AE, Honer WG, Falkai P. Hippocampal plasticity in response to exercise in schizophrenia. Arch Gen Psychiatry. 2010 Feb;67(2):133-43. doi: 10.1001/archgenpsychiatry.2009.193. PMID 20124113